CLINICAL TRIAL: NCT01355705
Title: A Phase 1 Study of Amrubicin in Combination With Lenalidomide and Weekly Dexamethasone in Relapsed/Refractory Multiple Myeloma
Brief Title: Phase 1-2 Amrubicin in Combo With Lenalidomide + Weekly Dexamethasone in Relapsed/Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Michaela Liedtke (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor-Investigator, Michaela Liedtke, Assistant Professor Medicine/Hematology, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-19092; AR_MM_PI_007 (Other: Celgene Corporation); SU-05062011-7711 (Other: Stanford University); HEMMYL0018 (Other: OnCore ID); IRB-19092 (Other: Stanford IRB)
Record Dates: First submitted 2011-05-16; First posted 2011-05-18 (Estimated); Results first posted 2017-03-03 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — amrubicin; Lenalidomide; Dexamethasone; Calcium Dobesilate; Aspirin; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Amrubicin + Lenalidomide + Dexamethasone (Experimental): Amrubicin will be given intravenously on Day 1 of each 3-week cycle beginning with 40 mg/m2, for a maximum of 4 cycles.
  Concurrent therapeutic medications:
  * Lenalidomide: 10 or 15 mg daily by mouth, Days 1 to 14
  * Dexamethasone: 40 mg weekly by mouth (Days 1, 8, and 15)
  Other drugs:
  * Aspirin: 81 or 325 mg daily oral
  * Pegfilgrastim subcutaneous on Day 2
  Interventions: Drug: Amrubicin; Drug: Lenalidomide; Drug: Dexamethasone; Drug: Aspirin; Drug: Pegfilgrastim

INTERVENTIONS:
Drug: Amrubicin — 40, 60, or 80 mg/m2 intravenous (IV)
  Other Names: SM-5887
Drug: Lenalidomide — 15 mg daily by mouth
  Other Names: CC-5013; Revlimid
Drug: Dexamethasone — 40 mg weekly by mouth
  Other Names: Decadron; Dexamethasone Intensol; Dexpak Taperpak
Drug: Aspirin — 81 or 325 mg daily by mouth
  Other Names: acetylsalicylic acid
Drug: Pegfilgrastim — 6 mg subcutaneous on Day 2
  Other Names: Neulasta; PEG-GCSF

SUMMARY:
To assess if amrubicin is safe and useful for patients with multiple myeloma requiring additional treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES

* Establish the maximum tolerated dose (MTD) and toxicity profile for the combination of amrubicin with lenalidomide and dexamethasone in previously treated adult patients with multiple myeloma during Phase I
* Determine the combined rate of complete response (CR) and very good partial response (VGPR) for this combination in this population as defined by the International Myeloma Working Group Uniform Response Criteria (IMWGURC)

SECONDARY OBJECTIVES

* Determine the overall response rate (CR, VGPR and PR)
* Assess additional evidence of ant-tumor activity as measured by duration of response (DOR), progression-free survival (PFS), time to tumor progression (TTP), and overall survival (OS)

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory multiple myeloma that has progressed following at least 1 prior therapy.
* Measurable disease defined as one of the following:

  * Serum M-protein ≥ 1 g/dL
  * Urine M-protein ≥ 200 mg/24 hours
* Received at least 1 prior line of systemic treatment that may have included lenalidomide and/or an anthracycline.
* No cytotoxic chemotherapy within 4 weeks prior to first dose of amrubicin. This interval may be reduced to 14 days for thalidomide, lenalidomide, bortezomib or corticosteroids, provided other entry criteria are met.
* Age ≥ 18 at the time of consent.
* Life expectancy of more than ≥ 3 months.
* No known central nervous system involvement by myeloma.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1 at study registration during phase 1. Once safety is confirmed, ECOG performance status 0 to 2 at study registration during phase 2.
* No poorly-controlled intercurrent illness.
* Platelets > 100 x 10^9/L
* Hemoglobin > 8.0g/dL
* Absolute neutrophil count (ANC) >1.5 x 10^9/L
* Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3 x upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 x ULN
* Calculated creatinine clearance ≥ 50 mL/min by Cockcroft-Gault formula.
* Left ventricular ejection fraction (LVEF) ≥ 50% by Echocardiogram (ECHO) or multiple gate acquisition scan (MUGA)
* All study participants must be registered into the mandatory RevAssist program, and be willing and able to comply with the Requirements of RevAssist.
* Disease-free of prior malignancies for ≥ 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast.
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 U/mL within 10 to 14 days and again within 24 hours prior to prescribing lenalidomide for Cycle 1 (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin 2 acceptable methods of birth control, one highly effective method and one additional effective method at the same time, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing.
* Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy.
* Ability to understand and the willingness to sign a written informed consent document.
* Able to adhere to the study visit schedule and other protocol requirements.
* Able to take aspirin (81 or ≥ 25 mg) daily as prophylactic anticoagulation. Patients intolerant to aspirin may use warfarin or low molecular weight heparin (LMWH). Patients with previous thromboembolic event on lenalidomide or thalidomide may be started on warfarin or LMWH. Patients already taking warfarin or LMWH do not require additional aspirin..
* Lactating females must agree not to breast-feed while taking lenalidomide

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Pregnant or breastfeeding females.
* Any concurrent severe or uncontrolled medical disease which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Use of any other experimental drug or therapy within 28 days of first dose of amrubicin.
* Known hypersensitivity to thalidomide or lenalidomide.
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
* LVEF ≤ 50%.
* Concurrent use of other anti-cancer agents or treatments.
* Known positive for HIV, or infectious hepatitis, type B or C.
* Cranial radiotherapy ≤ 21 days prior to first dose of amrubicin; radiotherapy to all other areas ≤ 7 days prior to first dose of amrubicin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michaela Liedtke, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dinner S, Dunn TJ, Price E, Coutre SE, Gotlib J, Berube C, Kaufman GP, Medeiros BC, Liedtke M. A phase I, open-label, dose-escalation study of amrubicin in combination with lenalidomide and weekly dexamethasone in previously treated adults with relapsed or refractory multiple myeloma. Int J Hematol. 2018 Sep;108(3):267-273. doi: 10.1007/s12185-018-2468-5. Epub 2018 May 25. PMID 29802551

RESULTS

PARTICIPANT FLOW:
Groups:
- Amrubicin + Lenalidomide + Dexamethasone: Amrubicin 40, 60, or 80 mg/m2 intravenous (IV) will be given intravenously on Day 1 of each 3-week cycle beginning with 40 mg/m2, for a maximum of 4 cycles.
  Concurrent therapeutic medications:
  * Lenalidomide: 10 or 15 mg daily by mouth, Days 1 to 14
  * Dexamethasone: 40 mg weekly by mouth (Days 1, 8, and 15)
  Other drugs:
  * Aspirin: 81 or 325 mg daily oral
  * Pegfilgrastim subcutaneous on Day 2
Period: Overall Study
Arm/Group | Amrubicin + Lenalidomide + Dexamethasone
Started | 14
Completed (1 subject completed but was not evaluable.) | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Amrubicin + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Response Rates After Amrubicin + Lenalidomide + Dexamethasone, Per International Myeloma Working Group Uniform Response Criteria
Description: Modified International Myeloma Working Group Uniform Response Criteria:
  Complete (CR)=
  * Negative for monoclonal protein (MP) in urine (U) and serum (S) +
  * No tissue plasmacytomas (PC) +
  * <5% plasma cells (PCs) in marrow (M)
  Stringent CR (sCR)= CR with normal light chain ratio+ no PCs in M
  Near CR (nCR)= CR, except MP persists in U and S
  Partial (PR)= S MP ≤50%, + U MP ≤90% or <200 mg/24 hours (hr)
  Very Good PR (VGPR)= in S MP ≤90%, + U MP <100 mg/24 hr
  Minimal (MR)=
  * S MP ≤51-75%, +
  * If light chain is excreted, reduced 50-89%/24 hr that is also >200 mg/24 hr, +
  * No increase in lytic bone lesions
  Progressive disease (PD)= any of:
  * S MP ≥125% and/or ≥+0.5 g/dL,
  * U MP ≥125% and/or ≥+200 mg/24 hr
  * New or increased bone lesions/PC
  * S calcium >11.5 mg/dL (attributed to increased PCs)
  PD after CR/sCR=
  * Reappearance of S or U MP
  * ≥5% clonal PCs in M
  * New PC, lytic bone lesions, hypercalcemia
  Stable Disease (SD)= Not CR, VGPR, MR, PR, or PD
Time Frame: 12 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Amrubicin + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 13
percentage of participants
  Complete Response (CR) rate | 0
  Very Good Partial Response (VGPR) Rate | 7.6
  Total CR + VGPR | 7.6
  Partial Response (PR) Rate | 15.4
  Overall Response Rate (ORR = CR + VGPR + PR) | 23

2. Secondary Outcome: Duration of Response (DOR)
Time Frame: 140 days
Measure: Median (Full Range); unit: days
Groups:
- Amrubicin + Lenalidomide + Dexamethasone: Amrubicin will be given intravenously on Day 1 of each 3-week cycle beginning with 40 mg/m2, for a maximum of 4 cycles.
  Concurrent therapeutic medications:
  * Lenalidomide: 10 or 15 mg daily by mouth, Days 1 to 14
  * Dexamethasone: 40 mg weekly by mouth (Days 1, 8, and 15)
  Other drugs:
  * Aspirin: 81 or 325 mg daily oral
  * Pegfilgrastim subcutaneous on Day 2
  Amrubicin: 40, 60, or 80 mg/m2 intravenous (IV)
  Lenalidomide: 15 mg daily by mouth
  Dexamethasone: 40 mg weekly by mouth
  Aspirin: 81 or 325 mg daily by mouth
  Pegfilgrastim: 6 mg subcutaneous on Day 2
Arm/Group | Amrubicin + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 13
days | 133 [129 to 140]

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) is alive and free from progression, per the modified International Myeloma Working Group Uniform Response Criteria, defined as any of:
  * Serum monoclonal protein ≥ 125% baseline and/or ≥ +0.5 g/dL from baseline,
  * Urine monoclonal protein ≥ 125% baseline and/or ≥ +200 mg/24 hour from baseline
  * New or increased bone lesions or plasmacytomas
  * Serum calcium > 11.5 mg/dL (attributed to increased plasma cells)
Time Frame: 9 months
Measure: Median (Full Range); unit: days
Arm/Group | Amrubicin + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 13
days | 96 [21 to 232]

4. Secondary Outcome: Time-to-next Treatment
Time Frame: 9 months
Measure: Median (Full Range); unit: days
Arm/Group | Amrubicin + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 13
days | 92 [24 to 281]

ADVERSE EVENTS:
Time Frame: Up to 12 weeks treatment, plus a minimum of 30 days follow-up
Arm/Group | Amrubicin + Lenalidomide + Dexamethasone
Serious Adverse Events (participants affected / at risk) | 3/14
Other Adverse Events (participants affected / at risk) | 12/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Amrubicin + Lenalidomide + Dexamethasone (N=14)
Sepsis (Infections and infestations) | 1
Cord compression (Nervous system disorders) | 1
Progressive disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — Hospitalization for infusional chemotherapy
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Amrubicin + Lenalidomide + Dexamethasone (N=14)
Thrombocytopenia (Blood and lymphatic system disorders) | 11
Anemia (Blood and lymphatic system disorders) | 12
Neutropenia (Blood and lymphatic system disorders) | 9
Deep venous thrombosis (Vascular disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 7
Anorexia (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 2
Elevated AST/ALT (Investigations) | 5
Hypoalbuminemia (Investigations) | 6
Infection (Infections and infestations) | 11
Insomnia (General disorders) | 2
Dysgeusia (General disorders) | 2
Headache (General disorders) | 1
Dizziness (Nervous system disorders) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 5
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Muscle cramps (Musculoskeletal and connective tissue disorders) | 2
Graft vs host diseae (GvHD) (Skin and subcutaneous tissue disorders) | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2
Creatinine (Investigations) | 4
Hypokalemia (Investigations) | 5
Fatigue (General disorders) | 7
Decreased ejection fraction (transient) (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No